CLINICAL TRIAL: NCT02557828
Title: Dynamic Need Tip Positioning With Ultrasound Versus Palpation Technique for Radial Artery Cannulation: A Prospective Randomized Controlled Trial
Brief Title: Target Sign vs Palpation for Radial Arterial Line Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator retired
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Roy K. Kiberenge, Associate- Physician, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 201505705
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Radial Artery Cannulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- palpation (Active Comparator): participants who are randomized to have radial arterial cannulation via palpation technique
  Interventions: Procedure: arterial line placement
- ultrasound (Active Comparator): participants who are randomized to have radial arterial cannulation via a new ultrasound technique
  Interventions: Procedure: arterial line placement

INTERVENTIONS:
Procedure: arterial line placement — radial arterial cannulation placed via palpation or ultrasound technique

SUMMARY:
Invasive blood pressure monitoring is achieved by cannulating an artery and transducing the pressure. During arterial cannulation the artery can be located by palpation, but use of ultrasound has increased the success rate of cannulation. A new ultrasound technique for vascular cannulation (dynamic needle tip positioning) has been described. Investigators aim to compare this technique to the palpation technique for arterial cannulation. Investigators hypothesize that the use of this novel ultrasound technique will result in a higher first attempt success rate and overall success compared to palpation.

Investigators plan to enroll 310 patients in this study. The participants in the study will have been deemed by the attending anesthesiologist to require a radial arterial line for the operation and thus the research protocol will not involve a deviation from the standard of care.

DETAILED DESCRIPTION:
Participants will be brought to the main operating rooms. The patient will not be required to do anything different than if they were not enrolled in the study. The anesthesiologist will be asked to confirm that the patient still requires an arterial line. The patient will be randomized either to palpation or ultrasound group. Patients would be placed in supine position on the operating room table and all regular monitors (electrocardiogram, pulse oximeter, non-invasive blood pressure) applied. After preoxygenation, the patient would be induced and the airway secured. For those requiring an arterial catheter before induction of general anesthesia, subcutaneous lidocaine will be used to anesthetize the planned puncture site.

The arms would be abducted and the decision on which side to place the arterial line will be determined by the operator after palpation or scanning the wrists with ultrasound. An ultrasound image of the radial artery to be cannulated will be obtained. A wrist roll would then be placed under the wrist and the hand secured with tape. The wrist would then be prepped with chlorhexidine and sterile towels placed around the prepped site. Timing would begin once the ultrasound or the operator fingers touch the prepped wrist. For those randomized to ultrasound, a Sonosite linear ultrasound probe would then be used to locate the radial artery. After satisfactory position is obtained, a 20 ga angiocath 45mm long would be used to puncture the artery and then would be advanced until the tip appears on the ultrasound view. When this happens the ultrasound is advanced about 2mm proximal along the artery. The needle is advanced until the tip is again visualized. This is repeated until the needle tip is in the lumen of the radial artery. At this point the needle is sequentially advanced in the lumen of the artery in small steps under ultrasound vision and then the cannula is advanced over the needle. The needle core is then retracted and the transducer is connected to the cannula. If the first attempt is unsuccessful, then more attempts may be made until 5 minutes elapse. Success is defined as arterial cannulation as shown by an arterial waveform that is obtained within 5 minutes of touching the prepped skin with an ultrasound probe or the operator fingers. After that the operator may use the arterial cannulation method of choice or decide to change to the other wrist.

For the palpation method, the radial artery would be palpated and then a 20 ga angiocath used to puncture the artery. After a return of blood in the catheter an attempt will be made to advance the catheter over the needle core. If this is not successful, the operator can make multiple attempts until 5 minutes elapse. After this time, the operator can use any desired method to cannulate the artery and may also decide to use the other wrist.

Investigators will record the successful first pass cannulation, and time to cannulate the vessel. Other measures will be number of attempts, number of catheters, radial artery depth, radial artery diameter, blood pressure, heart rate, and failure rate. Other data that will be recorded will include patient age, gender, weight, height , body mass index, and history of peripheral vascular disease, and diabetes.

Patients will not require any followup for the study.

ELIGIBILITY:
Inclusion Criteria:

* needing radial arterial cannulation intraoperatively

Exclusion Criteria:

* refusal to consent
* minors
* incarcerated individuals
* radial cannulation within past month
* negative modified Allen's test
* shock
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
first pass success | 5 minutes
  placement of arterial cannula in 5 minutes after touching the wrist

SECONDARY OUTCOMES:
overall success | 5 minutes
  successful arterial cannulation after any number of passes as long as it is within 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States